CLINICAL TRIAL: NCT04750031
Title: Evaluation of the Pain and Post Procedural Complications of Liver Biopsy Among Different Recovery Positions
Brief Title: Pain Scores and Complications do Not Differ at Three Recovery Position After Liver Biopsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Hasan Yılmaz, Assistant Professor, Kocaeli University
Other Study IDs: KouGasLVBx01
Record Dates: First submitted 2021-02-06; First posted 2021-02-11 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Pain, Acute; Liver Diseases
MeSH Terms: conditions — Acute Pain; Liver Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Liver Biopsy — Liver biopsy is a procedure to obtain small amount of liver by a needle.

SUMMARY:
Liver biopsy is still used as the gold standard in the diagnosis of many liver diseases. During the observation after liver biopsy, patients are hospitalized on their right side, which is the biopsy side, with the thought that adverse events (complications) such as bleeding or bile leakage will be less. Patients who do not develop complications after 4-6 hours of observation are discharged home. Some of the patients state that the right side-lying position for 4-6 hours is uncomfortable than the biopsy itself, and they prefer to lie on their back. In our study, researchers aim to investigate the rate of complications after biopsy, what recovery position found more acceptable by the patients.

DETAILED DESCRIPTION:
Liver biopsy is still used as the gold standard in the diagnosis of many liver diseases. The health practice notification (SUT) makes the diagnosis with liver biopsy mandatory for the treatment of chronic viral hepatitis (Chronic Hepatitis B Inf. And Chronic Hepatitis C Inf.). In daily gastroenterology practice, clinicians frequently perform a liver biopsy for the diagnosis of non-alcoholic fatty liver (NASH), and to a lesser extent, for the diagnosis of Wilson Disease and Hemochromatosis.

During the observation after liver biopsy, patients are hospitalized on their right side, which is the biopsy side, with the argument that there will be less bleeding or bile leakage complications. Patients who do not develop complications after 4-6 hours of observation are discharged to their homes. (1) In this study, researchers aimed to investigate the post-biopsy position of patients who were referred to the clinic for liver biopsy, the rate of complications after biopsy, and to what extent the patients found the procedure acceptable according to their post-biopsy position.

ELIGIBILITY:
Inclusion Criteria:

1. Cronic hepatitis B İnfection
2. Chronic hepatitis C İnfection
3. NASH
4. DILI
5. Acute or chronic liver damage caused unknown aetiology

Exclusion Criteria:

1.Refuse to give written informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute and chronic liver damaged patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Pain scores | Immediately after the procedure
  Patient reported pain scores will be assesed by visual analog scale, minimum score "0" refers no pain and "10" refers worst pain

SECONDARY OUTCOMES:
Complications | within 2 weeks after the procedure
  Complications such as liver lickage ,bleeding, infection at biopsy site will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University Medical Faculty Hospital, İzmit, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Anonymised pain scores and descriptive data
Supporting Information: CSR, Analytic Code
Time Frame: Data will be shared 3 months after the last patient recruited and it will be available 1 year.
Access Criteria: publicly aviable

REFERENCES:
- [Result] Costa RS, Cardoso AF, Ferreira A, Costa J, Costa D, Fernandes D, Caetano AC. What recovery position should patients adopt after percutaneous liver biopsy? Eur J Gastroenterol Hepatol. 2019 Feb;31(2):253-259. doi: 10.1097/MEG.0000000000001290. PMID 30358572